CLINICAL TRIAL: NCT06889675
Title: An Open-Label, Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of YB1-X7 Injection in Subjects with Advanced Solid Tumors
Brief Title: First in Human Study of YB1-X7 Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Salvectors Biotechnology LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZXK24-D1-P001
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Both administration routes will have three dose cohorts (low, medium, and high dose) , each cohort will have 3-6 subjects, following the standard 3+3 dose-escalation design, with single-dose multiple administrations in an escalating dose scheme.
  1. If no toxicities (DLTs ) in a dose cohort, the dose escalation study for the next dose cohort may proceed.
  2. If 1 of 3 subjects experience DLTs in the same dose cohort during the DLT observation period, 3 additional subjects will be enrolled in that dose cohort. If 0 of 3 newly enrolled msubjects experience DLTs, dose escalation may continue to the next cohort, if one or more DLTs occur among the newly enrolled three subjects, dose escalation will be stopped.
  3. If 2 of 3 or more subjects experience DLT, or 2 of 6 or more subjects experience DLT dose escalation will be stopped.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YB1-X7 Injection Intratumoral Injection (Experimental): YB1-X7 injection will be injected into the target lesion intratumorally. Three cohorts (low, medium, and high) will be assigned. The standard 3+3 dose-escalation design will be applied to explore dose limiting toxicity in 3 sequential cohorts with 3- 6 patients.
  Interventions: Drug: YB1-X7 Injection (IT)
- YB1-X7 Injection Intravenous Infusion (Experimental): YB1-X7 injection will be administered as an IV infusion through a dedicated line catheter over 2 hours.Three cohorts (low, medium, and high) will be assigned. The standard 3+3 dose-escalation design will be applied to explore dose limiting toxicity in 3 sequential cohorts with 3- 6 patients.
  Interventions: Drug: YB1-X7 Injection (IV)

INTERVENTIONS:
Drug: YB1-X7 Injection (IT) — Intratumoral injection
  Other Names: YB1-X7
  Arms: YB1-X7 Injection Intratumoral Injection
Drug: YB1-X7 Injection (IV) — Intravenous infusion
  Other Names: YB1-X7
  Arms: YB1-X7 Injection Intravenous Infusion

SUMMARY:
This clinical trial is an open-label, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetic, and preliminary efficacy of YB1-X7 injection in subjects with advanced solid tumors.

YB1-X7 injection is an attenuated Salmonella-based tumor therapy. It selectively accumulates in hypoxic tumor regions while being rapidly cleared from normal organs. After proliferating in the tumor microenvironment, YB1-X7 invades tumor cells and releases its therapeutic payload, leading to tumor cell death and tumor regression.

Conditions：To treat subjects with advanced and/or metastatic solid tumors who do not to respond to conventional standard treatment or who lack effective standard treatment.

DETAILED DESCRIPTION:
YB1-X7 is a genetically engineered attenuated Salmonella enterica strain. It has been further optimized based on the attenuated model of VNP20009 while inserting an anaerobic-targeting enrichment system, transforming YB1-X7 into a nutrient-deficient strain under aerobic conditions. This modification allows YB1-X7 to selective proliferation in hypoxic tumor regions while being cleared in normal oxygenated tissues, thereby achieving selective enrichment in tumor.

Additionally, YB1-X7 carries plasmids encoding the drug protein. Upon reaching the tumor region, YB1-X7 invades tumor cells, expressing and releasing drug protein, leading to tumor cell death and tumor regression.

This study is divided into two parts based on the route of administration:

Part 1: Subjects receiving intratumoral injection (IT). Part 2: Subjects receiving intravenous infusion (IV).

Both administration routes will have three dose cohorts (low, medium, and high dose) following the standard 3+3 dose-escalation design, with single-dose multiple administrations in an escalating dose scheme.

Each subject will receive only one administration method (IT or IV) and be assigned to only one dose cohort, completing the full treatment regimen for that dose level.

YB1-X7 injection will be administrated in 28-days cycles (once weekly for 3 weeks followed by 1-week rest).

For Subjects receiving intratumoral injection, superficial lesions can be injected directly, while deep-seated lesions may require ultrasound, CT, or endoscopic guidance for precise administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, no gender limitatlon
2. Subjects with advanced or metastatic solid tumors confirmed by pathological histology.
3. Subjects with advanced malignant solid tumors for whom standard treatment has failed or no other effective standard treatment available.
4. At least one measurable solid tumor by RECIST 1.1.
5. Subjects assigned to intratumoral injection must have at least one tumor that is suitable for biopsy or intratumoral injection.
6. Life expectancy must be at least 3 months.
7. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1.
8. Male and female subjects of childbearing potential should take effective contraceptive measures.

   ① Fertile women and men must agree to use acceptable contraceptive methods from the start of informed consent until at least 6 months after the last administration.
9. Laboratory blood test results during the screen period:

(1)No blood cell growth factors received within 14 days prior to testing.

① Absolute neutrophil count (ANC)≥1.5×109/L.

② Platelets≥90×109/L. Hemoglobin ≥90 g/L (blood transfusion is allowed to correct). (2) Serum albumin >30 g/L, total bilirubin <1.5×ULN, ALT and AST <2.5×ULN; for subjects with liver metastasis, ALT and AST <5×ULN; creatinine clearance ≥50 mL/min (Cockcroft-Gault formula) or Cr <1.5×ULN; (3) Prothrombin time (PT) and activated partial thromboplastin time (aPTT) <1.5×ULN.

10. Subjects understand the study and willing to sign the informed consent form.

Exclusion Criteria:

1.Pregnant or breastfeeding women. Subjects known to have a history of abuse of psychiatric drugs, alcoholism, or drug use.

3.Subjects who have previously undergone oncolytic bacteria treatment. 4.Subjects planning to surgery, radiation therapy, or other local treatments for target lesions during the study.

5.Subjects known to be allergic to the study drug or any of its excipients. 6.Subjects allergic or intolerant to antibiotics sensitive to Salmonella, such as amikacin cefpirome, ciprofloxacin,cefotaxime,meropenem.

7.Subjects currently using antibiotics. 8.Subjects who have not recovered fom adverse reactions of prior treatments (treatment-related toxicity grade≤2, except for hair loss, pigmentation, and other tolerable events determined by the investigator).

9.Subjects with active auto-immune diseases or prior diseases with recurrence potential (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroiditis.

10.Subjects with active or uncontrolled infections or unexplained fever≥38.5℃, including but not limited to bacterial infections, tuberculosis, herpes virus infections syphilis infections.

11.Subjects who underwent major surgery within 3 months prior to the first dose of the study drug (except for biopsies for diagnostic purposes).

12.Subjects who have received any anti-tumor treatment within 28 days or 5 half-lives prior to the first dose of the study drug, including chemotherapy, cell therapy, gene therapy, immunotherapy,biological agents, hormone therapy, targeted therapy, tumor drug embolization therapy.

13.Subjects who received radiation therapy within 28 days prior to the first dose of the study drug (except for local radiation therapy for pain relief).

14.Subjects who receive (live attenuated) virus vaccines: within 28 days prior to the first dose of the study drug, or during the study period or within 60 days after the last dose of the study drug.

Subjects who have used immunosuppressive drugs within 14 days prior to the first dose of the study drug (i.e., prednisone≥10 mg/day, dexamethasone≥1.5 mg/day), except for corticosteroid nasal sprays and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e., prednisone not exceeding 10 mg/day)or equivalent physiologica doses of other corticosteroids.

16. Subjects with known, uncontrolled, or symptomatic active central nervous system conditions.

17. Subjects with existing clinical symptoms or pooely controlled heart disease:

1. New York Heart Association (NYHA) class ≥II;
2. Unstable angina;
3. Myocardial infarction within the past year; Subjects with clinically significant supraventricular or ventricular arrhythmias needing treatment or intervention; Medicaion uncontrolled hypertension or hypotension (determined by the investigator); Subjects with valvular heart disease or mitral valve prolapse, aortic valve disease; Severe myocardial diseases. 18.Subjects known to have peripheral thromboembolic vascular diseases, aneurysms, or arterial/venous malformations.

19.Subjects Known allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

20.Subjects who are positive for Treponema pallidum antibodies, individuals with human immunodeficiency virus (HIV) infection, or known acquired immunodeficiency syndrome (AIDS).

21.Subjects with active hepatitis B (HBsAg positive and/or HBcAb positive with HBV-DNA ≥2000 IU/mL or requiring antiviral treatment), or those who test positive for hepatitis C virus (HCV) antibodies; or subjects co-infection with hepatitis B and C.

22.Other reasons unsuitable for the study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days post first dose.
  DLT is defined as any toxic reaction associated with the study drug occurring within 28 days after the first administration, graded refer to the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Adverse events (AEs) | From receiving study drug and throughout the study, until 28 days after the last dosing
  An AE is any untoward medical occurrence in a patient or clinical investigation patient, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Serious adverse events(SAEs) | From receiving study drug and throughout the study, until 28 days after the last dosing.
  A serious adverse event (SAE) refers to any medical event that results in:
  * Death
    * Life-threatening conditions ③ Permanent or severe disability or loss of function
      ④ Hospitalization or prolonged hospitalization
      ⑤ Congenital abnormalities or birth defects
  Other important medical events, which may not immediately threaten life, death, or require hospitalization, but still necessitate medical interventions to prevent one of the above outcomes, are also considered serious. Examples include:
  * Urgent treatments in an emergency room
    * Allergic bronchospasm (even if not requiring hospitalization) ③ Severe cachexia or seizures ④ Drug dependence or addiction Death due to drug-related adverse events (e.g., ventricular fibrillation) is classified as an SAE. However, if the death is due to the progression of the underlying disease (e.g., cancer) and the adverse event was mild (e.g., a rash or abdominal pain), it is not considered an SAE.

SECONDARY OUTCOMES:
YB1-X7 level in blood for PK analysis | Before the first administration up to 28 days after the last dosing.
  Evaluate the drug concentration and pharmacokinetics for subjects in different dose groups after the dose of either intratumoral injection or intravenous infusion.
Immunogenicity (anti-drug antibodies) | Before the first administration up to 28 days after the last dosing.
  The changes in the levels of anti-YB1-X7 antibodies (ADA) will be evaluated at different time points.
YB1-X7 level in blood for bacterial shedding. | Before the first administration up to 28 days after the last dosing.
  For subjects receiving intratumoral injection or intravenous infusion, blood samples will be collected in different dose groups.
YB1-X7 shedding level analysis in urine, saliva, faeces using qPCR | Before the first administration up to 28 days after the last dosing.
  For subjects receiving intratumoral injection or intravenous infusion, samples will be collected in different dose groups, including urine, saliva and faeces (or rectal swab), and the shedding level will be analysed using quantitative polymerase chain reaction (qPCR).
Cytokines | Before the first administration up to 28 days after the last dosing.
  Changes in cytokines in the blood at different time points. Cytokines including IFN-γ, IL-10, IL-12p70, IL-13, IL-1β, IL-2, IL-4, IL-6, IL-8, TNF-α.
Objective Response Rate (ORR) | From signing the informed consent form until 28 days after the last dose.
  ORR represents the proportion of subjects with complete or partial response, assessed using RECIST 1.1 criteria based on imaging.
Progression Free Survival (PFS) | From signing the informed consent form until 28 days after the last dose.
  PFS is defined as the time interval from date of first dose of YB1-X7 injection to the date of documented disease progression (iRECIST is used when the patient is suspected to be pseudo disease progression) or death due to any cause, whichever occurs first.
ime to Progression (TTP) | From signing the informed consent form until 28 days after the last dose.
  Time to Progression (TTP) is defined as the time from the start of treatment to the objective progression of the tumor.
Duration of Response (DOR) | From signing the informed consent form until 28 days after the last dose.
  Duration of Response (DOR) is defined as the time from the first assessment of Complete Response (CR) or Partial Response (PR) until Disease Progression (PD). It represents the duration that the tumor remains reduced following the treatment.
Overall Survival (OS) | 1 year
  OS will be evaluated for subjects in different dose groups who received intratumoral injection or intravenous infusion at Week 52 (1 year).
  Overall Survival (OS) is defined as the time from the start of treatment to death from any cause.
ECOG Performance Status Before and After Treatment | From baseline to week 12
  Changes in ECOG performance status will be assessed for subjects in different dose groups who received intratumoral injection or intravenous infusion compared to baseline.
  The score will refer to the Eastern Cooperative Oncology Group (ECOG) Performance Status.

IPD SHARING:
Plan to Share IPD: No
Due to confidentially and regulatory reasons